CLINICAL TRIAL: NCT00198107
Title: Novel Pharmacological Strategies in Autism
Brief Title: Evaluating the Effectiveness of Aripiprazole and D-Cycloserine to Treat Symptoms Associated With Autism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH072961 (NIH); R01MH072961 (NIH); DSIR 82-SEDR
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2019-03-29 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2018-04

CONDITIONS: Autistic Disorder
Keywords: Children; Adolescents; Aripiprazole; Cycloserine; Aggression; Irritability; Self-Injurious Behavior; Social Interaction; Antipsychotics; Pharmacology; Glutamatergic Agents
MeSH Terms: conditions — Autistic Disorder; Aggression; Self-Injurious Behavior | interventions — Aripiprazole; Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 Placebo (Placebo Comparator): Participants will take placebo
  Interventions: Drug: Placebo
- 2 Aripiprazole (Active Comparator): Participants will take aripiprazole
  Interventions: Drug: Aripiprazole
- 3 Aripiprazole + D-cycloserine (Active Comparator): Participants first will take aripiprazole then will also take D-cycloserine
  Interventions: Drug: Aripiprazole; Drug: D-cycloserine

INTERVENTIONS:
Drug: Aripiprazole — Participants will receive 8 weeks of initial treatment with aripiprazole. If responsive to treatment, participants may be assigned to an additional 16 weeks of aripiprazole and then an additional 8 more weeks of aripiprazole with D-cycloserine. Dosing schedule for participants less than 50 kg maximum dose will be 10 mg per day. Dosing schedule for participants greater than 50 kg maximum dose will be 15 mg.
  Other Names: Abilify
  Arms: 2 Aripiprazole; 3 Aripiprazole + D-cycloserine
Drug: Placebo — Participants assigned to placebo will take a placebo pill for the initial 8 weeks of treatment.
  Arms: 1 Placebo
Drug: D-cycloserine — D-cycloserine will be dosed in the range of 25 to 200 mg daily for the final 8 weeks of treatment.
  Arms: 3 Aripiprazole + D-cycloserine

SUMMARY:
This study will determine the effectiveness of aripiprazole and D-Cycloserine in treating symptoms associated with autism in children.

DETAILED DESCRIPTION:
Autism is a developmental disorder that affects every child differently. A wide range of symptoms accompany autism, including self-injurious behavior, aggression, and severe tantrums. Despite an improved ability to reduce these symptoms, existing drug treatments continue to be associated with adverse side effects. Also, there is no existing drug treatment that reliably improves social behavior, a core deficit in autism. Studies on drug treatment combinations that are designed to reduce self-injurious behavior, aggression, and severe tantrums and improve social behavior in children with autism have yet to be conducted. This study will address the above-mentioned limitations by evaluating aripiprazole in reducing self-injurious behavior, aggression, and severe tantrums and by evaluating the addition of D-Cycloserine in improving social behavior among children with autism.

This study will include three phases and an add-on component for some children. Participants will be randomly assigned to receive either aripiprazole or a placebo treatment for 8 weeks. Assessments measuring irritability, behavior, and social skills will be conducted at the end of this first phase. Those patients who respond well to aripiprazole will continue to receive aripiprazole treatment for another 16 weeks. This second phase will determine whether aripiprazole is associated with long-term maintenance of symptomatic improvement in patients who respond well to short-term treatment. Assessments will again be conducted at the end of this 16-week period. Those patients whose symptoms have stabilized and continue to improve while on aripiprazole will be asked to participate in the final phase of this study. During the this pilot phase, D-Cycloserine will be added to ongoing treatment with aripiprazole. Patients will take both aripiprazole and D-Cycloserine for an additional 8 weeks to determine if this combination of drug treatments results in improved social behavior once patients' aggression and self-injurious behavior have been stabilized with aripiprazole. At the end of this 8-week period, participants will be assessed for any changes in behavior, irritability, or social skills. Results from this study may aid in developing safer and more effective drug treatments for children and adolescents with autism.

ELIGIBILITY:
Inclusion Criteria:

* Weight of at least 15 kg (33.75 lbs)
* Meets DSM-IV criteria for autistic disorder
* Outpatient
* Medication-free for at least 2 weeks prior to baseline for all psychotropic medications. More information about this criterion, including exceptions, can be found in the protocol.
* Clinical Global Impression Scale Severity score (CGI-S) of at least 4
* Irritability subscale of the Aberrant Behavior Checklist (ABC) score of at least 18
* An IQ of at least 35 or a mental age of at least 18 months
* In good physical health

Exclusion Criteria:

* Meets DSM-IV criteria for Asperger's disorder, Rett's disorder, childhood disintegrative disorder, any other pervasive developmental disorder (PDD), schizophrenia, psychotic disorder, or bipolar disorder
* Current or past history of alcohol or other substance abuse within 6 months of study entry
* Comorbid neurodevelopmental disorder with possible association to autism (e.g., fragile-X syndrome, tuberous sclerosis)
* A significant medical condition such as heart, liver, kidney, or lung disease, or a seizure disorder
* Pregnant
* Prior adequate use of aripiprazole. More information about this criterion can be found in the protocol.
* Evidence of hypersensitivity to aripiprazole
* History of neuroleptic malignant syndrome

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2005-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J. McDougle, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Riley Hospital for Children, Christian Sarkine Autism Treatment Center, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711

RESULTS

PARTICIPANT FLOW:
Groups:
- 2 Aripiprazole: Participants will take aripiprazole
  Aripiprazole: Participants will receive 8 weeks of initial treatment with aripiprazole. If responsive to treatment, participants may be assigned to an additional 16 weeks of aripiprazole and then an additional 8 more weeks of aripiprazole with D-cycloserine. Dosing schedule for participants less than 50 mg maximum dose will be 10 mg per day. Dosing schedule for participants greater than 50 kg maximum dose will be 15 mg.
- 3 Aripiprazole + D-cycloserine: Participants first will take aripiprazole then will also take D-cycloserine
  Aripiprazole: Participants will receive 8 weeks of initial treatment with aripiprazole. If responsive to treatment, participants may be assigned to an additional 16 weeks of aripiprazole and then an additional 8 more weeks of aripiprazole with D-cycloserine. Dosing schedule for participants less than 50 mg maximum dose will be 10 mg per day. Dosing schedule for participants greater than 50 kg maximum dose will be 15 mg.
  D-cycloserine: D-cycloserine will be dosed in the range of 25 to 200 mg daily for the final 8 weeks of treatment.
Period: Double-Blind Period
Arm/Group | 1 Placebo | 2 Aripiprazole | 3 Aripiprazole + D-cycloserine
Started | 41 | 40 | 0
1 or More Follow-up Visits | 40 | 38 | 0
Completed | 35 | 37 | 0
Not Completed | 6 | 3 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Pilot Add-On Aripiprazole +D-cycloserine
Arm/Group | 1 Placebo | 2 Aripiprazole | 3 Aripiprazole + D-cycloserine
Started | 0 | 0 | 10
Completed | 0 | 0 | 8
Not Completed | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Placebo | 2 Aripiprazole | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41 | 40 | 81
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.4 (3.5) | 9.0 (2.9) | 9.2 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 34 | 36 | 70
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 40 | 81

OUTCOME MEASURES:

1. Primary Outcome: Mean Post-baseline Aberrant Behavior Checklist Irritability Score, Parent Report, Double-blind Phase
Description: The Aberrant Behavior Checklist (ABC) is a symptom checklist for assessing problem behaviors in individuals ages 6 to 54 with mental retardation. The full ABC is a 58-item parent rating with five factors: Irritability, Social Withdrawal, Stereotypy, Hyperactivity and Inappropriate Speech. It has been used as a primary outcome measure in several trials of children with developmental disabilities. The interpretation of the tool and its subscales is that higher scores, indicate greater severity. Fifteen item scores with values ranging from 0 (not a problem) to 3 (problem is severe) are summed to arrive at the total irritability scale store ranging from 0 to 45. Means were estimated using a repeated measures linear regression model with treatment group, baseline score, study week (in categories), and sex x Tanner stage stratum as covariates. A linear contrast estimated the average across study timepoints. Confidence intervals reflect a Bonferroni multiple testing correction accounting
Time Frame: Weeks 1, 2, 3, 4, 6, and 8
Population: All randomized study participants with at least one post-baseline ABC score. One participant assigned to placebo and 2 participants assigned to aripiprazole had no post-baseline assessments.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 1 Placebo | 2 Aripiprazole | 3 Aripiprazole + D-cycloserine
Number analyzed (Participants) | 40 | 38 | 0
units on a scale | 25.5 [22.8 to 28.3] | 18.6 [15.8 to 21.4] |

2. Primary Outcome: Odds of Improvement as Measured by the Clinical Global Impression-Global Improvement Scale (Improvement Defined as CGI-I=1 or CGI-I=2)
Description: Clinical Global Impressions (Guy, 1976) global improvement (CGI-I) is designed to take into account all factors to arrive at an assessment of response to treatment. The CGI-I scale ranges from 1 to 7, with lower scores indicating greater improvement (1=very much improved and 2=much improved). Participants with a CGI-I score of 1 or 2 were classified as improved. Odds were estimated using a repeated measures logistic regression model with treatment group, study week (in categories), and sex x Tanner stage stratum as covariates. A linear contrast estimated the average log odds across study timepoints. Confidence intervals reflect a Bonferroni multiple testing correction accounting for the selection of two primary outcomes.
Time Frame: Weeks 1, 2, 3, 4, 6 and 8
Population: All randomized study participants with at least one post-baseline CGI-I rating. One participant assigned to placebo and 2 participants assigned to aripiprazole had no post-baseline ratings.
Measure: Number (95% Confidence Interval); unit: odds
Arm/Group | 1 Placebo | 2 Aripiprazole | 3 Aripiprazole + D-cycloserine
Number analyzed (Participants) | 40 | 38 | 0
odds | 0.10 [0.05 to 0.23] | 0.50 [0.31 to 0.79] |

3. Secondary Outcome: Mean Post-baseline Aberrant Behavior Checklist Hyperactivity Score, Parent Report, Double-blind Phase
Description: The Aberrant Behavior Checklist (ABC) is a symptom checklist for assessing problem behaviors in individuals ages 6 to 54 with mental retardation. The full ABC is a 58-item Parent rating with five factors: Irritability, Social Withdrawal, Stereotypy, Hyperactivity and Inappropriate Speech. The 16-item Hyperactivity subscale covers overactivity, impulsiveness, inattention and noncompliance. It has been used as a primary outcome measure in several trials of children with developmental disabilities. The interpretation of the tool and its subscale is that higher scores, indicate greater severity. Sixteen item scores with values ranging from 0 (not a problem) to 3 (problem is severe) are summed to arrive at the total score ranging from 0 to 48. Means were estimated using a repeated measures linear regression model with treatment group, baseline score, study week (in categories), and sex x Tanner stage stratum as covariates. A linear contrast estimated the average across study timepoints.
Time Frame: Weeks 1, 2, 3, 4, 6 and 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 1 Placebo | 2 Aripiprazole | 3 Aripiprazole + D-cycloserine
Number analyzed (Participants) | 40 | 38 | 0
units on a scale | 29.7 [26.8 to 32.5] | 22.5 [19.6 to 25.4] |

4. Secondary Outcome: Mean Post-baseline Aberrant Behavior Checklist Inappropriate Speech Score, Parent Report, Double-blind Phase
Description: The Aberrant Behavior Checklist (ABC) is a symptom checklist for assessing problem behaviors in individuals ages 6 to 54 with mental retardation. The full ABC is a 58-item Parent rating with five factors: Irritability, Social Withdrawal, Stereotypy, Hyperactivity and Inappropriate Speech. It has been used as a primary outcome measure in several trials of children with developmental disabilities. The interpretation of the tool and its subscales is that higher scores, indicate greater severity. Four item scores with values ranging from 0 (not a problem) to 3 (problem is severe) are summed to arrive at the total inappropriate speech scale score ranging from 0 to 12. Means were estimated using a repeated measures linear regression model with treatment group, baseline score, study week (in categories), and sex x Tanner stage stratum as covariates. A linear contrast estimated the average across study timepoints.
Time Frame: Weeks 1, 2, 3, 4, 6, and 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 1 Placebo | 2 Aripiprazole | 3 Aripiprazole + D-cycloserine
Number analyzed (Participants) | 40 | 38 | 0
units on a scale | 7.4 [6.7 to 8.1] | 5.0 [4.2 to 5.7] |

5. Secondary Outcome: Mean Post-baseline Aberrant Behavior Checklist Social Withdrawal Score, Parent Report, Double-blind Phase
Description: The Aberrant Behavior Checklist (ABC) is a symptom checklist for assessing problem behaviors in individuals ages 6 to 54 with mental retardation. The full ABC is a 58-item Parent rating with five factors: Irritability, Social Withdrawal, Stereotypy, Hyperactivity and Inappropriate Speech. It has been used as a primary outcome measure in several trials of children with developmental disabilities. The interpretation of the tool and its subscales is that higher scores, indicates greater severity. Sixteen item scores with values ranging from 0 (not a problem) to 3 (problem is severe) are summed to arrive at the total social withdrawal scale score ranging from 0 to 48. Means were estimated using a repeated measures linear regression model with treatment group, baseline score, study week (in categories), and sex x Tanner stage stratum as covariates. A linear contrast estimated the average across study timepoints.
Time Frame: Weeks 1, 2, 3, 4, 6, and 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 1 Placebo | 2 Aripiprazole | 3 Aripiprazole + D-cycloserine
Number analyzed (Participants) | 40 | 38 | 0
units on a scale | 15.4 [13.4 to 17.5] | 11.7 [9.6 to 13.7] |

6. Secondary Outcome: Mean Post-baseline Aberrant Behavior Checklist Stereotypy Score, Parent Report, Double-blind Phase
Description: The Aberrant Behavior Checklist (ABC) is a symptom checklist for assessing problem behaviors in individuals ages 6 to 54 with mental retardation. The full ABC is a 58-item Parent rating with five factors: Irritability, Social Withdrawal, Stereotypy, Hyperactivity and Inappropriate Speech. It has been used as a primary outcome measure in several trials of children with developmental disabilities. The interpretation of the tool and its subscales is that higher scores, indicates greater severity. Seven item scores with values ranging from 0 (not a problem) to 3 (problem is severe) are summed to arrive at the total stereotypy scale score ranging from 0 to 21. Means were estimated using a repeated measures linear regression model with treatment group, baseline score, study week (in categories), and sex x Tanner stage stratum as covariates. A linear contrast estimated the average across study timepoints.
Time Frame: Weeks 1, 2, 3, 4, 6, and 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 1 Placebo | 2 Aripiprazole | 3 Aripiprazole + D-cycloserine
Number analyzed (Participants) | 40 | 38 | 0
units on a scale | 10.0 [8.9 to 11.1] | 7.2 [6.0 to 8.3] |

7. Secondary Outcome: Mean Post-baseline Score on a Modified Version of the Compulsion Subscale of the Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS)
Description: The CYBOCS- PDD is a semi-structured clinician-rated scale designed to rate the current severity of repetitive behavior in children with idiopathic autism spectrum disorders. Once the current repetitive behaviors are identified, they are rated on: Time Spent, Interference, Distress, Resistance, and Control. Each of these items is scored from 0 (least symptomatic) to 4 (most symptomatic), yielding a Total score from 0 to 20. Higher scores indicate higher severity. Means were estimated using a repeated measures linear regression model with treatment group, baseline score, study week (in categories), and sex x Tanner stage stratum as covariates. A linear contrast estimated the average across study timepoints.
Time Frame: Weeks 2, 4, 6 and 8
Population: All randomized study participants with at least one post-baseline CY-BOCS score. Two participants assigned to placebo and 2 participants assigned to aripiprazole had no post-baseline assessments.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 1 Placebo | 2 Aripiprazole | 3 Aripiprazole + D-cycloserine
Number analyzed (Participants) | 39 | 38 | 0
units on a scale | 14.4 [13.4 to 15.5] | 12.5 [11.5 to 13.5] |

8. Secondary Outcome: Mean Vineland Maladaptive Behavior Subscales Total Score, Week 8
Description: The Vineland Adaptive Behavior Scales, (Survey Interview Form) is a measure of adaptive behavior in children, adolescents and adults. It yields an overall standard score (Adaptive Behavior Composite, ABC) and age standard scores in four domains. ABC scores have a mean of 100 and a standard deviation of 15 (range = 20 to 160). Higher scores suggest a higher level of adaptive functioning. An increase in standard scores from Baseline to the Final Visit indicates improvement. Means were estimated using a repeated measures linear regression model with treatment group, study week (in categories, baseline or 8 weeks), and sex x Tanner stage stratum as covariates.
Time Frame: Week 8
Population: All randomized study participants. For 7 participants who exited the double-blind phase prior to week 8 but completed an exit interview (all assigned to placebo), week 8 scores were imputed using a last observation carried forward approach.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 1 Placebo | 2 Aripiprazole | 3 Aripiprazole + D-cycloserine
Number analyzed (Participants) | 41 | 40 | 0
units on a scale | 33.1 [29.6 to 36.6] | 23.1 [19.6 to 26.5] |

9. Secondary Outcome: Mean Autism Diagnostic Observation Schedule (ADOS) Social Affect and Restricted and Repetitive Behaviors Total Score, Week 8
Description: Autism Diagnostic Observation Scale (ADOS) (Lord), Modules 1-3 yields scores in 2 scales: Social Affect and Restricted and Repetitive Behavior. The ADOS has been repeatedly evaluated as a diagnostic measure, it has also been used as an outcome measure of autism severity (Aldred et al., 2004; Gutstein, 2007; Owly et al, 2001, Green et al, 2010). For modules 1-3, scores ranging from 0-2 on 14 items are summed to arrive at the Social Affect and Restricted and Repetitive Behavior Total Score, which ranges from 0 to 28. Higher scores indicate greater autism severity. Means were estimated using a repeated measures linear regression model with treatment group, study week (in categories, baseline or 8 weeks), and sex x Tanner stage stratum as covariates
Time Frame: Week 8
Population: All randomized study participants. For 9 participants who exited the double-blind phase prior to week 8 but completed an exit interview (8 assigned to placebo and 1 to aripiprazole), week 8 scores were imputed using a last observation carried forward approach.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 1 Placebo | 2 Aripiprazole | 3 Aripiprazole + D-cycloserine
Number analyzed (Participants) | 41 | 40 | 0
units on a scale | 19.0 [17.6 to 20.4] | 18.3 [17.0 to 19.7] |

10. Secondary Outcome: Mean Social Reciprocity Scale (SRS) Total Score, Week 8
Description: The 65-item SRS is a standardized measure of the core symptoms of autism. Each item is scored on a 4-point Likert scale. The score of each individual item is summed to create a total raw score. A total score results are as follows: 0-62: Within normal limits 63-79: Mild range of impairment 80-108: Moderate range of impairment 109-149: Severe range of impairment. Means were estimated using a repeated measures linear regression model with treatment group, study week (in categories, baseline or 8 weeks), and sex x Tanner stage stratum as covariates.
Time Frame: Week 8
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 1 Placebo | 2 Aripiprazole | 3 Aripiprazole + D-cycloserine
Number analyzed (Participants) | 41 | 40 | 0
units on a scale | 127.6 [119.8 to 135.3] | 112.6 [104.8 to 120.3] |

ADVERSE EVENTS:
Time Frame: Eight weeks or at the time of latest data collection.
Description: Adverse event information was collected via a structured side effect rating scale completed with the participant and their primary caregiver. This included a list of side-effects that have been reported with aripiprazole at a rate greater than 1%. The physician also asked about any visits to the doctor, new medication use, or any other complaints. Events that were not present at baseline and occurred or worsened after the date of randomization are reported.
Arm/Group | 1 Placebo | 2 Aripiprazole | 3 Aripiprazole + D-cycloserine
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/10
Other Adverse Events (participants affected / at risk) | 35/40 | 40/40 | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1 Placebo (N=40) | 2 Aripiprazole (N=40) | 3 Aripiprazole + D-cycloserine (N=10)
Change in Stool (Gastrointestinal disorders) | 2 | 2 | 0
Constipation (Gastrointestinal disorders) | 4 | 8 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 7 | 5
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Stomach or abdominal discomfort (Gastrointestinal disorders) | 4 | 7 | 2
Vomiting (Gastrointestinal disorders) | 8 | 15 | 3
Dry mouth (General disorders) | 2 | 2 | 0
Hypersalivation (General disorders) | 3 | 3 | 1
Appetite decrease (General disorders) | 6 | 12 | 1
Appetite increase (General disorders) | 11 | 16 | 3
Sedation/Drowsiness (General disorders) | 3 | 5 | 0
Tiredness/fatigue (General disorders) | 10 | 21 | 2
Fever (General disorders) | 2 | 3 | 0
Flu or upper respiratory problems (Infections and infestations) | 3 | 3 | 1
Nasal congestion or Cold (Infections and infestations) | 16 | 16 | 1
Weight gain (Metabolism and nutrition disorders) | 5 | 8 | 0
Weight loss (Metabolism and nutrition disorders) | 5 | 4 | 1
Headache (Nervous system disorders) | 8 | 3 | 1
Muscle rigidity (Nervous system disorders) | 0 | 3 | 0
Tremor (Nervous system disorders) | 0 | 3 | 0
Anxiety/Nervousness/Worry (Psychiatric disorders) | 0 | 3 | 1
Change in speech (Psychiatric disorders) | 7 | 3 | 2
Difficulty falling asleep (Psychiatric disorders) | 6 | 3 | 0
Increased motor activity (Psychiatric disorders) | 5 | 3 | 2
Increased repetitive speech (Psychiatric disorders) | 2 | 3 | 1
Interrupted sleep/other sleep problems (Psychiatric disorders) | 8 | 4 | 1
Irritability (Psychiatric disorders) | 7 | 3 | 2
Restlessness/Agitation, including fidgety (Psychiatric disorders) | 2 | 3 | 2
Sadness (Psychiatric disorders) | 0 | 3 | 0
Self-Injurious Behavior (Psychiatric disorders) | 1 | 3 | 0
Stereotypy (Psychiatric disorders) | 8 | 3 | 2
Enuresis (Renal and urinary disorders) | 2 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2
Localized rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 0
Dizziness/faintness (Vascular disorders) | 0 | 4 | 1
Intermittent nosebleed (Vascular disorders) | 0 | 3 | 0
Hypertalkativeness (Psychiatric disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No